CLINICAL TRIAL: NCT02280902
Title: Incidence and Risk Factors for Infections in Patient Treated With Corticosteroids, Immunosuppressive Drugs or Biotherapy for Immunologic and Inflammatory Diseases
Acronym: INFIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/25
Record Dates: First submitted 2014-09-19; First posted 2014-11-03 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Immunologic and Inflammatory Diseases
Keywords: auto-immune diseases; inflammatory diseases; risk factors; infections; cohort study
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — - Blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with immunologic and inflammatory diseases: Patient treated with corticosteroids, immunosuppressive drugs or biotherapy for immunologic and inflammatory diseases
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Systematic follow-up (M3, M6, M12, M18, M24, M30) will be implemented to complete epidemiologic, clinical, therapeutic and biological data during a 30 months period. Specific measure of immune cells, markers of immune activation, immunoglobulins as described above will be performed at M3, M6, M12 and M24. A biologic collection (serum and cells) will be performed at the same time points for future prognostic studies.

SUMMARY:
Infections represent the first cause of death and of morbidity in people treated for immunologic and inflammatory diseases with corticosteroids, immunosuppressive drugs or biotherapy. Epidemiological, clinical, biological and therapeutic determinants of these infections are poorly understood. There is no recommendation for the prevention and treatment of infections in this particular field.

Purpose : Recent therapeutic trials evaluating immunosuppressive and biotherapy (cyclophosphamide, mycophenolate mofetil, rituximab, belimumab) in the field of immunologic and inflammatory diseases have found a risk of severe infection of 7 to 18% during the first year after the beginning of the treatment. Thus, the main objective of the study is to describe the incidence and risk-factors for infections in people treated with such agents for immunologic and inflammatory diseases.

DETAILED DESCRIPTION:
Monitoring of neutrophils, lymphocytes, immune activation markers, immunoglobulins have not been prospectively studied in such patients. Preliminary retrospective studies have shown that total lymphopenia was independently associated with an increased risk of infections. A previous retrospective study from our group have also shown that total lymphopenia and CD3- lymphopenia three months after the beginning of rituximab was associated with infections.

The determinants of infections occurring during the course of immune and inflammatory diseases treated with corticoids and immunosuppressive drugs or biotherapy are probably multiples. We hypothesized that the following variables may have an impact on the risk of infections in those patients: Epidemiological: gender, social situation, Clinical: causal disease, comorbidities, vaccination status, Therapeutic: type and doses of corticosteroids and immunosuppressive drugs/biotherapy, prevention treatment Biological : neutrophils, total lymphocytes, CD4-T lymphocytes, CD8-T lymphocytes, B lymphocytes, immune activation (HLA-DR+ lymphocytes), CD5 and CD19 lymphocytes, CD27/IgD lymphocytes, immunoglobulins IgA, IgM, IgG.

On the other side, the impact of infection on the clinical course of immunologic or inflammatory disease have been poorly described and will be documented by this longitudinal study.

After inclusion in the present study, patients will be followed on a 30 months period and monitored at M3, M6, M12, M24 to describe the impact of treatment on clinical and biological variables. Every clinical event will be prospectively reported and validated by a specific committee.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Immune or inflammatory disease : Lupus, antiphospholipid syndrome, Sjogren syndrome, inflammatory myositis, immunologic thrombopenic purpura, autoimmune hemolytic anemia, Evan's syndrome, systemic vasculitis, Behcet disease.
* Indication of corticosteroid therapy > 20 mg for at least 3 months and/or immunosuppressive or biologic agent.
* Information consent

Exclusion Criteria:

* Previous treatment with immunosuppressive or biological agents, or cumulative dose of steroids > 1g last 6 months
* Splenectomy
* Pregnancy
* Evoluting Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated with corticosteroids, immunosuppressive drugs or biotherapy for immunologic and inflammatory diseases
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Viral, bacterila, fungal or parasitic infection leading to hospitalization | 30 months after the inclusion

SECONDARY OUTCOMES:
Biological and immunological markers | Each 6 months from baseline for 30 months
  The following items will be assessed every 6 months :
  total White blood cell CD3 CD4 CD8 HLA-DR+ B cells CD19+ B cells CD5+/- CD27/IgD NK cells IgA, IgM, IgG levels
Morbidity | Each 6 months from baseline for 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BONNET, Prof., Principal Investigator — University Hospital Bordeaux, France; Rodolphe THIEBAUT, Prof., Study Chair — University Hospital Bordeaux, France
Locations (7):
- France (7):
  - Service de Médecine Interne - CH d'Agen, Agen
  - Service de Médecine Interne et maladies Infectieuses - Hôpital Saint-André, Bordeaux
  - service de médecine interne - CH de Libourne, Libourne
  - Service de Médecine Interne - CHU de Limoges, Limoges
  - Service de Médecine Interne - CH de Pau, Pau
  - service Médecine Interne - CHU de Toulouse - Hôpital Purpan (5), Toulouse
  - service Médecine Interne - CHU de Toulouse - Hôpital Purpan (7), Toulouse